CLINICAL TRIAL: NCT02794376
Title: Mindfulness for Irritable Bowel Syndrome
Acronym: MIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11626
Record Dates: First submitted 2016-05-19; First posted 2016-06-09 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Mindfulness-Based Cognitive Therapy

ARMS (2):
- Immediate Treatment Group (Experimental): Mindfulness course consisting of six weekly two hour mindfulness sessions plus meditation homework assignments.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
- Delayed Treatment Group (Other): Waiting period plus Mindfulness course consisting of six weekly two hour mindfulness sessions plus meditation homework assignments after the waiting period has finished.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy (MBCT); Behavioral: Waiting Period

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
Behavioral: Waiting Period
  Arms: Delayed Treatment Group

SUMMARY:
This study investigates the effectiveness of a 6 week mindfulness intervention in reducing symptoms of Irritable Bowel Syndrome (IBS). All Participants will receive treatment. Participants will be randomly allocated to an immediate treatment group and a waiting list control group.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Diagnosed with IBS by Gastroenterologist or General Practioner (GP), meeting Rome III criteria for IBS, symptom onset at least 6 months prior to inclusion, discomfort or pain at least 2-3 days per month
* Participants speaks English fluently or at a native level
* Participant has normal or corrected to normal vision

Exclusion Criteria:

* Participant has insufficient manual dexterity for the computerized tasks
* Severe Diagnostic and Statistical Manual (DSM) Axis I or II psychiatric disorder (diagnosis of dementia, amnesia, delirium, a dissociative disorder, a personality disorder, schizophrenia or any other psychotic disorder, a substance-related or induced disorder (such as alcoholism), attention deficit hyperactivity disorder (ADHD), attention deficit disorder (ADD), primary diagnosis of obsessive compulsive disorder (OCD), current suicidality, regular non-suicidal self-injury.
* Recent bereavement (within one year)
* GI diagnosis other than IBS (IBD, coeliac disease, another FGID)
* Pregnancy
* No access to the internet
* Prior participation in an 8-week mindfulness course (MBSR, MBCT) or any other structured mindfulness training. Prior participation in Vipassana meditation courses. Regular meditation practice (meditating more than once per month).
* Not able or unwilling to commit to amount of practice (sessions and home practice).
* Participant is currently enrolled in another IBS treatment study (psychological or pharmacological).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Change in IBS symptom Severity (GSRS - IBS) | Baseline and Post Intervention (within the first three weeks of completion or the intervention)
  Self-Report Questionnaire

SECONDARY OUTCOMES:
Changes in IBS quality of Life (IBS-QOL) | Baseline and Post Intervention Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in Psychological Distress (DASS) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in Positive and Negative Emotions (PANAS) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in IBS catastrophizing (GI-Cognitions Questionniare) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in Visceral Anxiety Sensitivity (VSI) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in Mindfulness (FFMQ-short) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Self-Report Questionnaire
Changes in Attentional Control (ANT) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Behavioural Computer-based task
Changes in Illness Identification (IAT) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Behavioural Computer-based task
Changes in Shame Identification (IAT) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Behavioural Computer-based task
Changes in Attention to Health Threat (Dot-probe) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Behavioural Computer-based task
Changes in Shame Association (SRET) | Baseline and Post Intervention (within the first three weeks of completion or the intervention), Mid-Intervention (after 2 weeks of the start of the intervention)
  Behavioural Computer-based task
Change in IBS symptom Severity (GSRS - IBS) at Follow up | Baseline, Follow up (one month after the post assessment)
  Self-Report Questionnaire
Changes in IBS quality of Life (IBS-QOL) | Baseline, (Follow up one month after the post assessment)
  Self-Report Questionnaire
Baseline levels of Social Anxiety (SIAS-SPS) | Baseline
  Self-Report Questionnaire
Baseline levels of Alexithymia (TAS-20) | Baseline
  Self-Report Questionnaire
Baseline levels of Somatosensory Amplification (SSATS) | Baseline
  Self-Report Questionnaire
Baseline levels of Thought Suppression (WBSI) | Baseline
  Self-Report Questionnaire
Baseline levels of Rumination (RRS) | Baseline
  Self-Report Questionnaire

REFERENCES:
- [Derived] Henrich JF, Gjelsvik B, Surawy C, Evans E, Martin M. A randomized clinical trial of mindfulness-based cognitive therapy for women with irritable bowel syndrome-Effects and mechanisms. J Consult Clin Psychol. 2020 Apr;88(4):295-310. doi: 10.1037/ccp0000483. PMID 32134291